CLINICAL TRIAL: NCT04736537
Title: 4DCT Wrist Biomarkers During Resisted and Unresisted Tasks in Healthy Controls
Brief Title: A Study to Evaluate 4DCT Controls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Kristin Zhao, PhD, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-007668; R01AR071338 (NIH)
Record Dates: First submitted 2021-01-11; First posted 2021-02-03 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Wrist Ligament and Bone Disorders
MeSH Terms: conditions — Bone Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Healthy Controls (Experimental)
  Interventions: Device: 4DCT

INTERVENTIONS:
Device: 4DCT — CT imaging conceptually similar to time-lapse photography.

SUMMARY:
The purpose of this study is to use CT motion pictures (4DCT) to visualize and record how much space there is between certain wrist joint bones, both without any resistance and with light resistance to the movement, during a single scanning visit.

ELIGIBILITY:
Inclusion Criterion:

* Age ≥ 18 and ≤ 60 years.
* Control subjects without any history of wrist injury or disease.

Exclusion Criteria (applied to both wrists for control subjects):

* Previously-diagnosed rheumatological conditions or connective tissue diseases;
* Inability to be appropriately positioned in the scanner for the imaging;
* Congenital malformations of the wrist or forearm;
* Diagnosed wrist osteoarthritis
* Age under 18 or over 60.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin D. Zhao, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Controls
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Controls
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 24
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Scapholunate (SL) Gapping
Description: Normalized volar/dorsal location of the gapping at the scapholunate joint, measured in millimeters, at each of the 17 time steps during each movement.
Time Frame: Baseline
Measure: Median (Full Range); unit: millimeters
Arm/Group | Healthy Controls
Number analyzed (Participants) | 31
millimeters
  Radioulnar load, unresisted | 1.65 [1.15 to 2.52]
  Radioulnar load, resisted | 1.64 [1.24 to 2.54]
  Flexion-extension load, unresisted | 1.86 [1.29 to 3.30]
  Flexion-extension load, resisted | 1.92 [1.32 to 3.29]
  Grip load, unresisted | 1.83 [1.14 to 3.04]
  Grip load, resisted | 1.79 [0.97 to 2.95]

2. Primary Outcome: Radioscaphoid (RS) Gapping
Description: Normalized volar/dorsal location of the gapping at the radioscaphoid joint, measured in millimeters, at each of the 17 time steps during each movement.
Time Frame: Baseline
Measure: Median (Full Range); unit: millimeters
Arm/Group | Healthy Controls
Number analyzed (Participants) | 31
millimeters
  Radioulnar load, unresisted | 1.42 [-0.49 to 2.04]
  Radioulnar load, resisted | 1.39 [-1.15 to 1.72]
  Flexion-extension, unresisted | 1.52 [0.59 to 1.96]
  Flexion-extension, resisted | 1.50 [0.95 to 1.75]
  Grip load, unresisted | 1.48 [0.82 to 1.83]
  Grip load, resisted | 1.49 [0.89 to 1.80]

3. Primary Outcome: Radiolunate (RL) Gapping
Description: Normalized volar/dorsal location of the gapping at the radiolunate joint, measured in millimeters, at each of the 17 time steps during each movement.
Time Frame: Baseline
Measure: Median (Full Range); unit: millimeters
Arm/Group | Healthy Controls
Number analyzed (Participants) | 31
millimeters
  Radioulnar load, unresisted | 1.81 [0.28 to 2.03]
  radioulnar load, resisted | 1.88 [1.29 to 2.06]
  Flexion-extension load, unresisted | 1.56 [0.39 to 2.18]
  Flexion-extension load, resisted | 1.79 [1.19 to 2.05]
  Grip load, unresisted | 1.77 [1.36 to 2.12]
  Grip load, resisted | 1.76 [1.49 to 2.16]

4. Secondary Outcome: Scaphotrapezium (STm) Gapping
Description: Normalized volar/dorsal location of the gapping at the scaphotrapezium joint, measured in millimeters, at each of the 17 time steps during each movement.
Time Frame: Baseline
Measure: Median (Full Range); unit: millimeters
Arm/Group | Healthy Controls
Number analyzed (Participants) | 31
millimeters
  Radioulnar load, unresisted | 1.06 [0.83 to 1.65]
  Radioulnar load, resisted | 1.13 [0.84 to 1.66]
  Flexion-extension load, unresisted | 1.18 [0.65 to 1.75]
  Flexion-extension load, resisted | 1.13 [0.75 to 1.56]
  Grip load, unresisted | 1.14 [0.77 to 1.71]
  Grip load, resisted | 1.10 [0.75 to 1.68]

5. Secondary Outcome: Scaphotrapezoid (STd) Gapping
Description: Normalized volar/dorsal location of the gapping at the scaphotrapezoid joint, measured in millimeters, at each of the 17 time steps during each movement.
Time Frame: Baseline
Measure: Median (Full Range); unit: millimeters
Arm/Group | Healthy Controls
Number analyzed (Participants) | 31
millimeters
  Radioulnar load, unresisted | 0.97 [0.79 to 1.66]
  Radioulnar load, resisted | 1.04 [0.62 to 1.59]
  Flexion-extension load, unresisted | 1.09 [0.61 to 1.39]
  Flexion-extension load, resisted | 1.09 [0.57 to 1.37]
  Grip load, unresisted | 1.26 [0.55 to 1.62]
  Grip load, resisted | 1.19 [0.42 to 1.51]

6. Secondary Outcome: Trapezoitrapezoid (TmTd) Gapping
Description: Normalized volar/dorsal location of the gapping at the trapeziotrapezoid joint, measured in millimeters, at each of the 17 time steps during each movement.
Time Frame: Baseline
Measure: Median (Full Range); unit: millimeters
Arm/Group | Healthy Controls
Number analyzed (Participants) | 31
millimeters
  Radioulnar load, unresisted | 0.52 [0.32 to 0.78]
  Radioulnar load, resisted | 0.55 [0.32 to 0.77]
  Flexion-extension load, unresisted | 0.54 [0.34 to 0.83]
  Flexion-extension load, resisted | 0.54 [0.36 to 0.79]
  Grip load, unresisted | 0.54 [0.31 to 0.75]
  Grip load, resisted | 0.55 [0.30 to 0.73]

ADVERSE EVENTS:
Time Frame: Single scanning visit, approximately 30 minutes.
Arm/Group | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT04736537/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/37/NCT04736537/ICF_001.pdf